CLINICAL TRIAL: NCT04111705
Title: A Phase II Non-randomized, Single Group Assignment, Open-label, Multicenter Study of Efficacy and Safety of Lorlatinib Monotherapy After Failure of First-line Second-generation ALK Kinase Inhibitor in Patients With Advanced ALK-positive Non-small Cell Lung Cancer
Brief Title: Lorlatinib After Failure of First-line Second-generation ALK Kinase Inhibitor in Patients With Advanced ALK-positive Non-small Cell Lung Cancer
Acronym: ORAKLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1902
Record Dates: First submitted 2019-08-30; First posted 2019-10-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: IFCT; ORAKLE; NSCLC; ALK-positive; monotherapy
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: A phase II non-randomized, single group assignment, open-label, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lorlatinib (Experimental): 100 mg once daily
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — 100 mg once daily

SUMMARY:
Crizotinib is a first-generation ALK tyrosine kinase inhibitor (ITK-ALK). It is the standard first-line treatment for patients with advanced NSCLC with ALK gene rearrangement. Alectinib, ceritinib and brigatinib are second-generation ITK-ALK. They have been shown to be effective in the first line of treatment in randomized trials. Alectinib has shown superiority to crizotinib as the first line of treatment in three randomized therapeutic trials, positioning this ITK-ALK as the treatment of choice in first-line treatment. Despite the effectiveness of these new treatments, all patients will virtually experience a relapse. There is no data on second-generation TKI-ALK resistance mechanisms when given as first-line treatment and the best therapeutic strategy for progression is undefined.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent:

   * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing
2. Patients with histologically or cytologically confirmed locally advanced not eligible to a local treatment or metastatic NSCLC (Stage IIIB or IV accordingly to 8th classification TNM, UICC 2015) that carries an ALK rearrangement, as determined by the molecular biology platform of the investigator by FISH assay or by Immunohistochemistry (IHC), or Next Generation Sequencing (NGS) or RNA sequencing approach .
3. Disease Status Requirements: Disease progression meeting RECISTv1.1 after first-line alectinib or brigatinib only. No prior chemotherapy is allowed in the metastatic disease setting.
4. Tumor Requirements: All Patients must have at least one measurable target lesion according to RECIST v1.1. In addition, patients with asymptomatic and neurologically stable CNS metastases (including patients controlled with stable or decreasing steroid use within the last week prior to study entry) will be eligible. The brain metastases may be newly diagnosed after disease progression with alectinib or brigatinib or be present as progressive disease after surgery, whole brain radiotherapy or stereotactic radiosurgery (see Exclusion Criterion for the lapsed time period required between the end of radiotherapy and study entry). Patients who have leptomeningeal disease (LM) or carcinomatous meningitis (CM) will be eligible if the LM/CM is visualized on MRI or if documented baseline cerebral spinal fluid (CSF) positive cytology is available and asymptomatic and neurologically stable (including patients controlled with stable or decreasing steroid use within the last week prior to study entry).
5. Tumor Sample Requirement: Tumour biopsy sampling on fresh tissue (FFPE blocks required) at time of progression on first-line TKI is mandatory. Tumour biopsy should be exploitable for molecular analysis. If the tumour biopsy is not exploitable, the inclusion will be allowed if two blood samples are provided for tumoral cfDNA analysis. The Sponsor will monitor a posteriori the exploitability of provided tumour biopsies and will investigate the impossibility to perform or repeat tissue tumor sampling.
6. Age ≥18 years.
7. Life expectancy of at least 12 weeks, in the opinion of the Investigator.
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2
9. Adequate Bone Marrow Function, including:

   * Absolute Neutrophil Count (ANC) ≥1.5 x 109/L;
   * Platelets ≥100 x 109/L;
   * Hemoglobin ≥9 g/dL.
10. Adequate Pancreatic Function, including:

    * Serum lipase ≤1.5 x ULN.
11. Adequate Renal Function, including:

    * Serum creatinine ≤1.5 x ULN or estimated creatinine clearance ≥60 mL/min as calculated using the method standard for the institution.
12. Adequate Liver Function, including:

    * Total serum bilirubin ≤1.5 x ULN;
    * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN; ≤5.0 x ULN if there is liver metastases involvement.
13. Participants must have recovered from treatment toxicities to CTCAE Grade ≤ 1 (for participants who have developed interstitial lung disease [ILD], they must have fully recovered) except for AEs that in the investigator' judgment do not constitute a safety risk for the patient.
14. Participants must have recovered from effects of any major surgery, or significant traumatic injury, at least 35 days before the first dose of lorlatinib
15. For all females of childbearing potential, a negative pregnancy test must be obtained within the screening period. A patient is of childbearing potential if, in the opinion of the investigator, she is biologically capable of having children and is sexually active. Additionally, all females of childbearing potential must provide an agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 90 days after the last dose of study drug.
16. For men: agreement to remain abstinent or use a barrier method of contraception (e.g., condom) during the treatment period and for at least 90 days after the last dose of study drug and agreement to refrain from donating sperm during this same period.
17. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
18. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedure.
19. Participant has national health insurance coverage.
20. Washout period: if previous progression on ALK-TKI: 7 days from last dose of the drug. The washout period may be shortened to 2 days at investigator discretion.

Exclusion Criteria:

1. Patients who experienced a clinical benefit of less than 6 months with front-line alectinib or brigatinib.
2. Participants with disease progression on front-line treatment with 2G ALK-TKI i.e. brigatinib or alectinib limited to CNS or one non-CNS site (oligometastasis) and eligible to a local ablative treatment (surgery or stereotaxic radiotherapy).
3. Transdifferentiation into small cell lung cancer.
4. Spinal cord compression is excluded unless the patient demonstrates good pain control attained through therapy and there is stabilization or recovery of neurological function for the 4 weeks prior to study entry.
5. Patients with symptomatic and neurologically instable CNS metastases or leptomeningeal metastasis (including patients that require increasing doses of steroids within one week prior to Day 0 of screening phase and during the screening phase to manage CNS symptoms).
6. Major surgery within 35 days of study entry. Minor surgical procedures (eg, port insertion, mediastinoscopy, surgical procedure for re-sampling) are not excluded, but sufficient time at investigator discretion should have passed for wound healing.
7. Radiation therapy within 2 weeks of study entry (except palliative to relieve bone pain). Palliative radiation (≤15 fractions) must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have completed at least 2 weeks prior to study entry. Whole brain radiation must have completed at least 4 weeks prior to study entry.
8. Prior therapy with an antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including, but not limited to, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4.
9. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
10. Clinically significant cardiovascular disease (that is, active or <3 months prior to enrollment): cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec.
11. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, athletic patients etc.), machine-read ECG with QTc >470 msec, or congenital long QT syndrome.
12. Patients with predisposing characteristics for acute pancreatitis according to investigator judgment (eg, uncontrolled hyperglycemia, current gallstone disease, alcoholism [more than 4 drinks on any day or 14 drinks per week where 1 drink is defined as the alcoholic beverage containing approximately 14 grams of pure alcohol, eg, 12 fl oz/360 mL regular beer or 5 fl oz/150 mL of wine] in the last month.
13. History of bilateral or Grade 3 or 4 interstitial fibrosis or diffuse interstitial lung disease. Patients with history of prior radiation pneumonitis are not excluded.
14. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
15. Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, DCIS of the breast or localized and presumed cured prostate cancer) within the last 3 years.
16. Active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease or previous gastric resection or lap band.
17. Current use or anticipated need for food or drugs prohibited (see chapter 8.9.2 for details).
18. Patients presenting with abnormal Left Ventricular Ejection Fraction (LVEF) by echocardiogram or Multi-Gated Acquisition Scan (MUGA) according to institutional lower limits.
19. Breastfeeding female patients (including patients who intend to interrupt breastfeeding).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the Objective Response Rate (ORR) at 6 weeks. | Time from enrollment until 6 weeks after treatment.
  ORR is defined as the proportion of patients achieving an objective response (complete response (CR) or partial response (PR)) according to Response Evaluation Criteria in Solid Tumors (RECIST), v.1.1 (RECIST 1.1), as assessed by the investigators.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) assessed by an independent review committee (IRC). | Time from enrollment until 6 weeks after treatment
  Response according to RECIST v.1.1 as assessed by an independent review committee (IRC)
PFS in overall population and in cohort A, B and C. | Approximately 8 months after randomization
  PFS is defined as the time between the date of inclusion and the first date of documented disease progression according to RECIST 1.1 as assessed by the investigator and the IRC or death from any cause during the study, whichever occurs first.
Disease Control Rate (DCR) in overall population and in cohort A, B and C. | Percentage of participants with CR, PR, or stable disease (SD) for at least twelve weeks (according to RECIST 1.1)
  DCR is defined as the percentage of participants with CR, PR, or stable disease (SD) for at least twelve weeks, according to RECIST 1.1.
Duration of Response (DOR) in overall population and in cohort A, B and C. | Approximately 1 year
  DOR is defined as the time from the first occurrence of an objective response (CR or PR), based on RECIST 1.1 to first documented disease progression or death assessed by an IRC.
Overall Survival . | Approximately 1 year
  OS is defined as the time from the first lorlatinib dose and death from any cause during the study. OS will be assessed at 6 months, at 12 months and at 18 months.
Time to Tumor Response (TTR). | Approximately 1 year
  TTR is defined as the time from the first lorlatinib dose and the first occurrence of an objective response (CR or PR) based on RECIST 1.1 and assessed by an IRC.
Central Nervous System (CNS) ORR. | Approximately 1 year
  CNS ORR is defined as the proportion of patients achieving an objective response (complete response (CR) or partial response (PR)) of the baseline measurable and non-measurable CNS disease according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria, as assessed by an IRC.
CNS PFS. | Approximately 1 year
  CNS PFS is defined as the proportion of patients achieving an objective response (complete response (CR) or partial response (PR)) of the baseline measurable and non-measurable CNS disease according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria, as assessed by an IRC
CNS DOR. | Approximately 1 year
  CNS DOR is defined as the time from the first occurrence of an objective response (CR or PR) of the baseline measurable and non-measurable CNS disease for at least twelve weeks, according to RECIST 1.1. and Revised Assessment in Neuro Oncology (RANO) criteria, as assessed by an IRC.
CNS TTR. | Approximately 1 year
  CNS TTR is defined as the time from the first lorlatinib dose and the first occurrence of an objective response (CR or PR) of the baseline measurable and non-measurable CNS disease, according to RECIST 1.1. and Revised Assessment in Neuro Oncology (RANO) criteria, as assessed by an IRC.
Best ORR and PFS depending on prior brigatinib or alectinib treatment | Approximately 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Duruisseaux, Study Chair — Lyon - URCOT; Denis Moro-Sibilot, Study Chair — Grenoble - CHU
Locations (32):
- France (32):
  - Angers - CHU, Angers
  - Annecy - CH, Annecy
  - Bayonne - CH, Bayonne
  - Besançon - CHU, Besançon
  - Bordeaux - CHU Hôpital Haut-Lévèque, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne-Billancourt
  - Caen - CHU Côte de Nacre, Caen
  - Colmar - CH, Colmar
  - Créteil - CHI, Créteil
  - Dijon - CRLCC, Dijon
  - Grenoble - CHU, Grenoble
  - Le Mans - CHG, Le Mans
  - Lille - Hôpital Calmette, Lille
  - Lyon - CRLCC, Lyon
  - Marseille - AP-HM Hôpital Nord, Marseille
  - Marseille - Institut Paoli Calmette, Marseille
  - Montpellier - CHU, Montpellier
  - Montpellier - Clinique, Montpellier
  - Mulhouse - GHRMSA, Mulhouse
  - Nantes - CRLCC, Nantes
  - Orléans - CHR, Orléans
  - Paris - APHP - Hopital Tenon, Paris
  - Paris - APHP Bichat, Paris
  - Paris - Curie, Paris
  - Paris - Hôpital Cochin, Paris
  - Lyon - URCOT, Pierre-Bénite
  - Saint Quentin - CH, Saint-Quentin
  - Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Toulon - CHI, Toulon
  - Toulouse - CHU, Toulouse
  - Vandoeuvre-lès-Nancy - CRLCC, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/488-ifct-1902